CLINICAL TRIAL: NCT00820898
Title: A Phase II Evaluation of Gemcitabine (Gemzar®, LY188011) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Gemcitabine in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0129Q; NCI-2009-01175 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0129Q; CDR0000631591; GOG-0129Q (Other: Gynecologic Oncology Group); GOG-0129Q (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2015-05

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Recurrent Uterine Corpus Carcinoma
MeSH Terms: interventions — Gemcitabine

ARMS (1):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011

SUMMARY:
This phase II trial is studying the side effects of gemcitabine and to see how well it works in treating patients with recurrent or persistent endometrial cancer. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the antitumor activity of gemcitabine hydrochloride in patients with persistent or recurrent endometrial adenocarcinoma who have failed higher priority treatment protocols.

II. To determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial adenocarcinoma

  * Recurrent or persistent disease
  * Refractory to curative therapy or established treatments
* The following epithelial cell types are eligible:

  * Endometrioid adenocarcinoma
  * Serous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Adenocarcinoma not otherwise specified
  * Mucinous adenocarcinoma
  * Squamous cell carcinoma
  * Transitional cell carcinoma
  * Mesonephric carcinoma
* Measurable disease, defined as ≥1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR as ≥ 10 mm by spiral CT scan
* Must have ≥ 1 target lesion

  * Tumors within a previously irradiated field are designated as target lesions provided there is documented disease progression or biopsy confirmed persistent disease ≥ 90 days after completion of radiotherapy
* Must have received 1 prior chemotherapeutic regimen for management of endometrial cancer

  * Initial treatment may have included non-cytotoxic agents or high-dose therapy, consolidation therapy, or extended therapy administered after surgical or non-surgical assessment

    * No more than one prior cytotoxic chemotherapy regimen (either with single or combination cytotoxic drug therapy)

      * One additional non-cytotoxic regimen for management of recurrent or persistent disease is allowed
* Not eligible for a higher priority GOG protocol, if one exists (i.e., any active Phase III GOG protocol for the same patient population)
* GOG performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No neuropathy (sensory and motor) > grade 1, according to NCI CTCAE v3.0
* No active infection requiring antibiotics (except an uncomplicated urinary tract infection)
* No other invasive malignancies within the past 5 years except non-melanoma skin cancer
* No prior cancer treatment that contraindicates study therapy
* Recovered from prior surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy for endometrial cancer
* At least 3 weeks since prior biological therapy, immunotherapy, or other therapy for endometrial cancer
* At least 4 weeks since prior radiotherapy
* More than 3 years since prior radiotherapy for localized breast cancer, head and neck cancer, or skin cancer and

  * No recurrent or persistent breast cancer, head and neck cancer, or skin cancer
* More than 3 years since prior adjuvant chemotherapy for localized breast cancer

  * No recurrent or metastatic breast cancer
* No prior radiotherapy to any portion of the abdominal cavity or pelvis except for the treatment of endometrial cancer
* No prior chemotherapy for any abdominal or pelvic tumor except for the treatment of endometrial cancer
* No prior gemcitabine hydrochloride

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tait, Principal Investigator — Gynecologic Oncology Group
Locations (20):
- United States (20):
  - Hartford Hospital, Hartford, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Gynecologic Oncology Group, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Zale Lipshy University Hospital, Dallas, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on February 2, 2009 and was closed to accrual on July 27, 2009.
Groups:
- Gemcitabine: Gemcitabine 800mg/m2 I.V. Days 1 and 8 every 21 days (one cycle)
Period: Overall Study
Arm/Group | Gemcitabine
Started | 24
Completed (Eligible and treated patients) | 23
Not Completed | 1
Not completed — Inelgible - wrong primary site | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Gemcitabine
Number analyzed (Participants) | 23
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1
  50-59 years | 8
  60-69 years | 8
  70-79 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine
Number analyzed (Participants) | 23
Participants
  Partial response | 1
  Complete response | 0

2. Primary Outcome: Incidence of Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Participants
  Leukopenia | 6 | 6 | 8 | 3 | 0 | 0
  Thrombocytopenia | 5 | 11 | 5 | 1 | 1 | 0
  Neutropenia | 10 | 1 | 7 | 4 | 1 | 0
  Anemia | 5 | 6 | 7 | 4 | 1 | 0
  Hemorrhage | 22 | 1 | 0 | 0 | 0 | 0
  Nausea/Vomiting | 14 | 6 | 3 | 0 | 0 | 0
  Gastrointestinal | 7 | 7 | 8 | 1 | 0 | 0
  Alopecia | 19 | 2 | 2 | 0 | 0 | 0
  Dermatologic | 21 | 0 | 2 | 0 | 0 | 0
  Renal | 20 | 1 | 1 | 0 | 1 | 0
  Alkaline Phosphatase | 20 | 3 | 0 | 0 | 0 | 0
  SGOT | 20 | 2 | 1 | 0 | 0 | 0
  Neurotoxicity | 14 | 8 | 1 | 0 | 0 | 0
  Constitutional | 6 | 10 | 6 | 1 | 0 | 0
  Metabolic | 18 | 2 | 2 | 1 | 0 | 0
  Pulmonary | 17 | 2 | 1 | 0 | 1 | 2
  Lymphatics | 21 | 1 | 0 | 1 | 0 | 0
  Infection | 20 | 0 | 2 | 1 | 0 | 0
  Pain | 17 | 5 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Gemcitabine
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=23)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1
Pain: Abdominal Pain Nos (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Renal Failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (N=23)
Neutrophils (Blood and lymphatic system disorders) | 16
Platelets (Blood and lymphatic system disorders) | 20
Leukocytes (Blood and lymphatic system disorders) | 18
Lymphopenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 22
Pulmonary Hypertension (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Inr (Vascular disorders) | 1
Ptt (Vascular disorders) | 1
Sweating (General disorders) | 1
Weight Gain (General disorders) | 1
Fever (General disorders) | 6
Weight Loss (General disorders) | 2
Rigors/Chills (General disorders) | 1
Fatigue (General disorders) | 19
Insomnia (General disorders) | 3
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 5
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Heartburn (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dentures (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Anorexia (Gastrointestinal disorders) | 5
Dehydration (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Limb (Blood and lymphatic system disorders) | 8
Ast (Metabolism and nutrition disorders) | 3
Gfr (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Ggt (Metabolism and nutrition disorders) | 1
Alt (Metabolism and nutrition disorders) | 3
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 1
Mood Alteration - Anxiety (Nervous system disorders) | 2
Cognitive Disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Neuropathy-Sensory (Nervous system disorders) | 10
Blurred Vision (Eye disorders) | 1
Pain: Urethra (General disorders) | 2
Pain: Chest Wall (General disorders) | 1
Pain: Head/Headache (General disorders) | 1
Pain: Neck (General disorders) | 1
Pain: Extremity-Limb (General disorders) | 2
Pain: Back (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 7
Pain: Skin (General disorders) | 1
Pain: Middle Ear (General disorders) | 1
Pain: Muscle (General disorders) | 3
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Urinary Frequency (Renal and urinary disorders) | 3
Flu-Like Syndrome (General disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less